CLINICAL TRIAL: NCT07044440
Title: The Development and Evaluation of a Digital Follow-up Program During the Initial Four Weeks After Discharge Home Following Thoracic Surgery. A Confirmatory, Single-center, Prospective, Non-blinded, Randomized, Controlled Study
Brief Title: Digital Follow-up Program After Discharge Home Following Thoracic Surgery
Acronym: DFP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-00796;kt25Lardinois3
Record Dates: First submitted 2025-06-16; First posted 2025-07-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Thoracic Surgery; Mobile Health; Post Operative Recovery; Follow-up
Keywords: Electronic Follow-up; Thoracic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital follow-up (Experimental): digital follow-up by questionnaire in addition to routine follow-up
  Interventions: Other: digital outpatient follow-up
- standard follow-up (Active Comparator): routine follow-up
  Interventions: Other: standard follow-up

INTERVENTIONS:
Other: digital outpatient follow-up — In addition to routine outpatient follow-up visits on day 14 and 28 post-operative, digital follow-up by questionnaire on their health status and general well-being are provided. Possibility to request an interaction with a doctor from our department at any time during the 28 days following discharge
  Arms: digital follow-up
Other: standard follow-up — routine outpatient follow-up visits on day 14 and 28 post-operative
  Arms: standard follow-up

SUMMARY:
The aim of the study is to evaluate whether a digital follow-up program can improve postoperative pain management and quality of life in patients during the first 28 days after discharge home following thoracic surgery, compared to standard follow-up care.

DETAILED DESCRIPTION:
Thoracic surgery is essential for treating conditions such as thoracic malignancies, trauma, and chronic pulmonary diseases. While often life-saving, recovery after thoracic surgery can be challenging. Enhanced Recovery After Surgery (ERAS) programs have improved outcomes across surgical fields, but their impact on postoperative quality of life (QoL) in thoracic surgery is under-researched.

QoL post-surgery involves factors such as pain, physical and respiratory function, psychological well-being, and return to daily life. Effective communication between patients and their physicians post-discharge is crucial for early detection and management of complications.

Studies in other surgical areas (e.g., colorectal and cardiac surgery) have shown that mobile apps for follow-up can reduce emergency visits, readmissions, and improve patient experience. However, similar evidence is scarce in thoracic surgery. Existing studies suggest electronic patient-reported outcome (ePRO) systems could help monitor symptoms and improve care, but further research is needed.

Despite promising results in other specialties, there is limited evidence on the use of digital tools to monitor and support recovery after thoracic surgery. Given the importance of pain management, QoL, and preventing complications, the researchers aim to explore whether a digital follow-up program could offer measurable benefits for patients recovering at home.

The study aims to develop and evaluate a digital follow-up program for patients in the first 28 days after discharge home from thoracic surgery. The primary objective is to assess whether active, digital patient-physician communication can improve postoperative pain outcomes, compared to standard follow-up care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed an informed consent form and underwent a surgery performed at the Thoracic Surgery Department of the University Hospital Basel
* Age ≥ 18 years at the time of informed consent
* First participation in the Study
* Patient operated under general anesthesia
* Patients who are in possession of a smart phone or personal computer and have an e-mail account and are able to answer a digital questionnaire. Or an immediate caretaker in the same household owns a smartphone or personal computer and is familiar with the use
* Patients who understand verbal and written German or French
* Patients discharged at home after surgery
* Hospital stay > 3 nights after surgery

Exclusion Criteria:

* Patients under preoperative opioid/cortisone therapy
* Patients who are unable to follow the procedure of the study, e. g. read or understand German or French, psychological disorders, dementia, etc.
* Enrolment of the investigator, his/her family members, employees and other dependent person
* Patients with polytrauma or who underwent mediastinoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Subjective pain perception | 4 weeks after discharge home
  Impact on the subjective pain perception is assessed by the numeric rating scale (NRS). Scale ranges from 0-10 while 10 indicates more pain

SECONDARY OUTCOMES:
General well-being | 4 weeks after discharge home
  General well-being is assessed by the numeric rating scale (NRS). Scale ranges from 0-10 while 10 indicates better outcome
Post-Discharge documentation of analgesic use | During the 4 weeks after discharge home
  Assessment of any analgesics admitted after discharge home
Emergency consultations | During the 4 weeks after discharge home
  Number of emergency consultations within 4 weeks after discharge home
Readmissions | During the 4 weeks after discharge home
postoperative complications | During the 4 weeks after discharge home
  postoperative complications after hospital discharge home according to the Clavien-Dindo Classification of surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: Didier Lardinois, Prof. MD, Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland